CLINICAL TRIAL: NCT07386041
Title: Lung Ultrasound-Guided Respiratory Management in Infants: A Single-Center Randomized Controlled Trial
Brief Title: Lung Ultrasound-Guided Respiratory Management in Infants
Acronym: NeoLUS-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006737
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Respiratory Failure

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1 ratio to either the lung ultrasound-guided respiratory management group or the standard care group. Both groups are followed concurrently to compare outcomes.
Who Masked: Outcomes Assessor
Masking Description: Clinical care teams cannot be blinded due to the nature of the intervention. Outcome assessors and statisticians analyzing study outcomes will remain blinded to group assignment. Therefore it will be single masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Lung ultrasound guided respiratory management (Experimental): Participants randomized to this group will under lung ultrasound assessments at predefined clinical time points. Lung ultrasound scores will guide:
  * Surfactant administration in the early neonatal period
  * Weaning from non-invasive respiratory suppport
  * Transition to room air
  Decisions will follow predefined lung ultrasound score thresholds using a validating scoring system. Ultrasounds to be performed by trained neonatal providers using standardized techniques. Attending neonatologists may override protocol recommendations if clinically necessary, with documentation
  Interventions: Procedure: Lung ultrasound-guided respiratory management
- Control - Standard Clinical Care (No Intervention): Participants randomized to this group will receive respiratory management based on standard NICU clinical criteria including oxygen requirement, work of breathing, blood gas measurements, and radiographic findings. Lung ultrasound may be performed if clinically indicated, but will not be used for protocolized decision making.

INTERVENTIONS:
Procedure: Lung ultrasound-guided respiratory management — Scheduled lung ultrasounds are performed to guide decisions about surfactant administration, non-invasive respiratory support weaning, and transition to room air using predefined lung ultrasound score thresholds.
  Arms: Intervention - Lung ultrasound guided respiratory management

SUMMARY:
This single-center randomized controlled study will compare lung ultrasound-guided respiratory management with standard clinical care in infants requiring respiratory support.

The primary outcome measure is length of NICU stay.

DETAILED DESCRIPTION:
Infants, especially premature infants, frequently require respiratory support in the neonatal intensive care unit (NICU). Lung ultrasound is a bedside, radiation-free tool that can assess lung aeration and guide respiratory management, but its effect on clinical outcomes has not been evaluated in a U.S. randomized trial.

This single-center randomized controlled study will compare lung ultrasound-guided respiratory management with standard clinical care in premature infants requiring respiratory support. In the intervention group, lung ultrasound scores will guide surfactant administration, weaning non-invasive respiratory support, and weaning from non-invasive respiratory support to room air using predefined thresholds. The control group will use standard care to guide surfactant administration, weaning non-invasive respiratory support, and weaning from non-invasive respiratory support to room air.

The primary outcome is length of NICU stay. Secondary outcomes include duration of respiratory support, time on non-invasive respiratory support, time to successful weaning to room air, need for re-intubation, surfactant dosing, and mortality prior to discharge. This study aims to determine whether lung ultrasound-guided management can improve respiratory care and reducive hospital length of stay in infants requiring respiratory suppport.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the Tufts Medical Center NICU
* Requiring invasive or non-invasive respiratory support
* Requiring surfactant therapy
* Parental or guardian informed consent obtained

Exclusion Criteria:

* Major congenital anomalies
* Known chromosomal abnormalities
* Congenital diaphragmatic hernia
* Decision for comfort care
* Surfactant administered prior to transfer from outside hospital (only excluded for surfactant decisions)

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Length of NICU stay (days) | From date of NICU admission to date of hospital discharge up to one year

SECONDARY OUTCOMES:
Duration of any respiratory support | From date of initiation of respiratory support to date of discontinuation of respiratory support, up to one year
Duration of non-invasive respiratory support | From date of initiation of non-invasive respiratory support to date of discontinuation of non-invasive respiratory support up to one year.
Time to successful weaning to room air | From date of initiation of respiratory support to date of sustained room air without support for at least 48h, up to one year.
Weaning failure | From date of weaning respiratory support, to date of re-escalation of respiratory support if needed, up to 72 hours
Need for reintubation | From date of extubation, to date of reintubation, up to 72 hours.
Number of surfactant doses administered | Number of surfactant doses quantified over the course through study completion, up to an average of 1 year.
Mortality prior to discharge | From date of birth until the date of death from any cause, assessed up to one year.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung Ultrasonography Score to Evaluate Oxygenation and Surfactant Need in Neonates Treated With Continuous Positive Airway Pressure. JAMA Pediatr. 2015 Aug;169(8):e151797. doi: 10.1001/jamapediatrics.2015.1797. Epub 2015 Aug 3. PMID 26237465
- [Background] Gathright M, Chacko A, Paulson M, O'Connor B, Mansky R, Lasarev M, Cowan E, Hulse W, Monroe E, Alfaro E, Baker M, Bauer AS, Diego E. An Evaluation of Vital Signs in Intubated Neonates Undergoing Lung Point-of-Care Ultrasound in the Neonatal Intensive Care Unit. J Clin Ultrasound. 2025 Dec 22. doi: 10.1002/jcu.70161. Online ahead of print. PMID 41427513